CLINICAL TRIAL: NCT04554563
Title: The Effect of Core Stability Training on the Transverse Abdomen and Multifidus Muscles Morphology in Young Non-specific Low Back Pain Individuals.
Brief Title: The Effect of Core Stability Training on Deep Stabilizing Muscles.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Responsible Party: Principal Investigator, Tomasz Kuligowski, PHD., Assistant Professor, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USG TrA MF
Record Dates: First submitted 2020-09-12; First posted 2020-09-18 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Low Back Pain, Mechanical; Low Back Pain; Low Back Pain, Postural
Keywords: low back pain; ultrasound; sonofeedback; core stability; lumbar spine; transverse abdomen; multifidus
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): 4-week core stability training
  Interventions: Other: Core stability training
- Control group (No Intervention): Standard physical therapy

INTERVENTIONS:
Other: Core stability training — 20 sessions of specific core stability exercise with no external loading.
  Arms: Training group

SUMMARY:
Non-specific low back pain is the most cause of adult disability throughout life. Its prevalence widens in young adults. Background of this pathology can be multifactorial. One of the most common is poor core stability and overloading of the local tissues as a result.

Among treatment methods stabilizing training is commonly used with good effects. This form of therapy affects the transverse abdomen and multifidus muscles. To assess these structures several methods can be applied, e.g. sonofeedback.

Our hypothesis claims that the core muscles morphology will change over the training process duration, in result, the analgesic effect will be achieved.

DETAILED DESCRIPTION:
Non-specific low back pain is the most cause of adult disability throughout life. Its prevalence widens in young adults. Background of this pathology can be multifactorial. One of the most common is poor core stability and overloading of the local tissues as a result.

Among treatment methods stabilizing training is commonly used with good effects. This form of therapy affects the transverse abdomen (TrA) and multifidus (MF) muscles. To assess these structures several methods can be applied, e.g. sonofeedback.

All participants will be randomly divided into two groups:

1. Training group (TG)
2. Control group (CG)

Outcome measure:

Pre- and post-therapy outcome measure will be done. It will include:

* ultrasound (sonofeedback) of the TrA and MF
* Oswestry Disability Index questionnaire (ODI)
* subjective pain scale - Numeric Rating Scale (NRS)

Intervention:

Core stability training including 4 exercise positions, each of 15 repetitions, 4 sets. Once a day, 5 times a week, 20 sessions in total (4 weeks).

Our hypothesis claims that the core muscles morphology will change over the training process duration, in result, the analgesic effect will be achieved.

ELIGIBILITY:
Inclusion Criteria:

* low back pain
* age from 18 to 30 years old
* written consent of the participants

Exclusion Criteria:

* injuries of the spine
* fractures of the spine
* surgery interventions in the spine region prior to the study
* psychiatric disorders
* neurologic disorders

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Ultrasound | 5 minutes
  Non-invasive measure of the TrA and MF muscles
Pain level | 1 minute
  Numeric Rating Scale. Picking the number on a scale from 0 to 10.
Questionnaire | 5 minutes
  Oswestry Disability Index questionnaire - subjective disability measure throughout daily living activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinika Fizjoterapii, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Masse-Alarie H, Beaulieu LD, Preuss R, Schneider C. Repetitive peripheral magnetic neurostimulation of multifidus muscles combined with motor training influences spine motor control and chronic low back pain. Clin Neurophysiol. 2017 Mar;128(3):442-453. doi: 10.1016/j.clinph.2016.12.020. Epub 2016 Dec 28. PMID 28160750
- [Background] Hides JA, Walsh JC, Smith MMF, Mendis MD. Self-Managed Exercises, Fitness and Strength Training, and Multifidus Muscle Size in Elite Footballers. J Athl Train. 2017 Jul;52(7):649-655. doi: 10.4085/1062-6050-52.3.13. Epub 2017 May 1. PMID 28459281
- [Background] Finta R, Nagy E, Bender T. The effect of diaphragm training on lumbar stabilizer muscles: a new concept for improving segmental stability in the case of low back pain. J Pain Res. 2018 Nov 28;11:3031-3045. doi: 10.2147/JPR.S181610. eCollection 2018. PMID 30568484